CLINICAL TRIAL: NCT03151057
Title: Idelalisib Post Allogeneic Hematopoietic Stem Cell Transplant (HSCT) in B Cell Derived Malignancies: A Phase 1 Double Blinded Randomized Placebo Toxicity Trial
Brief Title: Idelalisib Post Allogeneic Hematopoietic Stem Cell Transplant (HSCT) in B Cell Derived Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety endpointreached
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J1633; IRB00157704 (Other: JHMIRB)
Record Dates: First submitted 2017-03-29; First posted 2017-05-12 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: B Cells-Tumors; B Cell Chronic Lymphocytic Leukemia; Follicular Lymphoma; Mantle Cell Lymphoma; Large B-Cell Diffuse Lymphoma of Bone (Diagnosis)
Keywords: Idelalisib; Zydelig; allo transplant; PI3K inhibitor; post transplant maintenance therapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Disease | interventions — idelalisib

STUDY DESIGN:
Intervention Model Description: Idelalisib 100mg or placebo twice daily, starting day +90 (+-/ 10 days) after transplant until day +270.
Who Masked: Participant, Investigator
Masking Description: Participant, investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Idelalisib 100mg (Experimental): Idelalisib is an orally-administered, selective inhibitor of Phosphoinositide 3 kinase (PI3K)-delta which has been shown to be extremely effective in inducing partial to complete responses in many B-cell derived malignancies.
  intervention: 100mg Idelalisib twice daily beginning +90(+/- 10) days after allo HSCT and continued through Day 270 post transplant
  Interventions: Drug: Idelalisib 100 MG
- Placebo oral tablet (Placebo Comparator): Placebo to be taken twice daily beginning +90(+/- 10) days after allo HSCT and continued through Day 270 post transplant
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Idelalisib 100 MG — 100mg BID beginning on day 90 (+/- 10days) and continuing until day 270 post transplant.
  Other Names: Zydelig
  Arms: Idelalisib 100mg
Drug: Placebo Oral Tablet — placebo
  Arms: Placebo oral tablet

SUMMARY:
This is a study to evaluate the safety of idelalisib as post-transplantation maintenance in patients with B cell hematologic malignancies undergoing a allogeneic hematopoietic stem cell transplant (HSCT). Safety will be evaluated through the assessment of cytopenias, effect on donor chimerism, effect on the incidence and severity of acute graft versus host disease, and gastro-intestinal tolerance.

DETAILED DESCRIPTION:
Currently, to improve overall survival, the focus of the BMT program at JHH the introduction of anti-neoplastic therapy post transplantation: where the allo BMT serves as a platform to allowing a new intolerant immune system to interact with the post allo BMT intervention.

The importance of post BMT therapy has been made evident with tyrosine kinase inhibition (TKI) in Philadelphia chromosome positive acute lymphocytic leukemia (ALL) and chronic myeloid leukemia(CML), where patients who had disease progression while on TKI therapy pre-allo BMT enjoy marked improvement in overall survival when TKI is part of a maintenance program; the use of DNA hypomethylation agents after allo BMT for relapsed myeloid malignances; or the use of rituximab after allo BMT in follicular lymphoma.

Idelalisib, an orally-administered, selective inhibitor of Phosphoinositide 3 kinase (PI3K), is extremely effective in inducing partial responses to complete responses in many B-cell derived malignancies and should be studied in the post alloHSCT setting. Johns Hopkins Hospital has one of the world's largest experiences with alloHSCT. This study proposes a double blinded randomized phase I placebo trial where all patients who have undergone alloHSCT for a B-cell derived hematologic malignancy be offered either idelalisib 100mg or placebo twice daily for 180 days starting approximately 90 days after their HSCT.

ELIGIBILITY:
INCLUSION CRITERIA

1. >18 years of age
2. Has undergone allo HSCT to treat a B-cell derived hematologic malignancy: accepted alloHSCT regimens include: myeloablative or reduced intensity conditioning from any donor (matched, partially mismatched or cord) and any source (peripheral blood, bone marrow, or cord).
3. T bili ≤ 1.5 mg/dL except for patients with Gilbert's syndrome or hemolysis
4. AST, ALT and alk phos all < 2.5X ULN
5. Karnofsky performance score ≥ 40
6. ECOG ≤3
7. For women of childbearing potential, a negative serum or urine pregnancy test with sensitivity less than 50 mIU/m within 72 hours before the start of study medication.
8. Use of two forms of contraception with less than a 5% failure rate or abstinence by all transplanted patients for a minimum of 1 month after the last dose of Idelalisib. For the first 60 days post-transplant, transplant recipients should be encouraged to use non-hormonal contraceptives due to the potential adverse effect of hormones on bone marrow engraftment.
9. Ability to receive oral medication.
10. Ability to understand and provide informed consent.

EXCLUSION CRITERIA

1. ECOG >3 (Karnofsky <40%)
2. ALT, AST >2.5 ULN or total bilirubin >1.5 ULN (not attributable to Gilbert's)
3. Women who are pregnant or breastfeeding.
4. Exclude if patient has cirrhosis or is currently being actively treated for hepatitis C.
5. History of positive HIV-1 or HIV-2 serologies or nucleic acid test.
6. Active hepatitis B infection as documented by positive Hepatitis B PCR assay
7. Use of investigational drug, other than the study medications specified by the protocol, within 30 days of transplantation.
8. Receipt of a live vaccine within 30 days of receipt of study therapy.
9. ≥ Grade II aGVHD
10. The presence of any medical condition that the Investigator deems incompatible with participation in the trial
11. Subjects who are required to use a medication classified as a strong CYP3A inducer of inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Gladstone, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double blinded randomized study with 2 participants randomized to idelalisib arm for every 1 randomized to placebo.
Groups:
- Idelalisib 100mg: Idelalisib is an orally-administered, selective inhibitor of Phosphoinositide 3 kinase (PI3K)-delta which has been shown to be extremely effective in inducing partial to complete responses in many B-cell derived malignancies.
  intervention: 100mg Idelalisib twice daily beginning +90(+/- 10) days after allo HSCT and continued through Day 270 post transplant
  Idelalisib 100 MG: 100mg BID beginning on day 90 (+/- 10days) and continuing until day 270 post transplant.
Period: Overall Study
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 57.33 [28 to 71] | 58.00 [49 to 69] | 57.62 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 4 | 10
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Treatment-limiting Toxicities Will be Defined as Idelalisib Interruption for >14 Days, or Other >3 Adverse Events as Defined by CTCAE IV Not Captured in the Protocol for Dose De-escalation.
Description: The evaluation of the safety of Idelalisib as post-transplantation maintenance in patients with B cell hematologic malignancies
Time Frame: Day 90 - Day 270 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

2. Secondary Outcome: Event Free Survival at One Year.
Description: Impact of Idelalisib on aGVHD, relapse, and non-relapse mortality
Time Frame: Beginning Day 90 post transplant until Day 360
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

3. Secondary Outcome: Identify Potential Predictive Biomarker Candidates Based on Exploratory Gene Expression Analysis of Immune Biomarkers in Bone Marrow Aspirates and Whole or Targeted Exome Sequencing of Lymphoma Cells
Description: Search for Biomarkers which could better identify which patients would respond to treatment with Idelalisib in the post-transplant setting.
Time Frame: Beginning Day 90 post transplant until Day 270
Population: Exploratory gene expression analysis of immune biomarkers in bone marrow aspirates and whole or targeted exome sequencing of lymphoma cells was not was not performed on any samples for this study. This study was terminated early due to safety concerns. Samples collected were not analyzed due to an initial lack of lab staffing during COVID then were destroyed after this sponsor/investigator left Johns Hopkins.
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 17 months
Arm/Group | Idelalisib 100mg | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 2/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/9 | 4/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib 100mg (N=9) | Placebo Oral Tablet (N=7)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0) — CMV viremia
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 4 (4) | 1 (1) — neutropenia
diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
increased Alanine transaminase (ALT) (Investigations) | 2 (3) | 2 (2) — increased Alanine transaminase increased at least 3x upper limit of normal value.
Increased Aspartate Transferase (AST) (Investigations) | 2 (2) | 2 (2) — Aspartate Transferase (AST) increased at least 3x upper limit of normal value.
Increased bilirubin (Investigations) | 1 (1) | 0 (0) — Bilirubin increased at least 3x upper limit of normal
sepsis (Infections and infestations) | 0 (0) | 1 (1) — Systemic bacterial infection
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhagic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
Decreased platelet count (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idelalisib 100mg (N=9) | Placebo Oral Tablet (N=7)
idelalisib or placebo held for >14 days (General disorders) | 5 (5) | 3 (3)
Graft versus host disease (GVHD) (Immune system disorders) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT03151057/Prot_SAP_000.pdf